CLINICAL TRIAL: NCT05305443
Title: COVID-19 Treatment Cascade Optimization Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Comprehensive Behavioral Health Center (Unknown); North Jersey Community Research Initiative (Other); University of Michigan (Other)
Responsible Party: Principal Investigator, Liliane Cambraia Windsor, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: UIUC-IRB 22606; 1U01AI169469-01 (NIH)
Record Dates: First submitted 2022-03-30; First posted 2022-03-31 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: SMART Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Navigation/tested/navigation services (Experimental): After initial randomization, some participants will be assigned to receive navigation services(NS). Those who complete the COVID-19 testing will again be randomized and some will continue receiving NS.
  Interventions: Behavioral: Navigation Services
- Navigation/tested/brief counseling (Experimental): After initial randomization, some participants will be assigned to receive navigation services (NS). Those who complete the COVID-19 testing will again be randomized and some will be assigned to receive Brief Counseling (BC)
  Interventions: Behavioral: Navigation Services; Behavioral: Brief Counseling
- Navigation/not tested/navigation services (Experimental): After initial randomization, some participants will be assigned to receive navigation services (NS). Those who do not complete the COVID-19 testing will again be randomized and some will continue receiving NS.
  Interventions: Behavioral: Navigation Services
- Navigation/not tested/critical dialogue (Experimental): After initial randomization, some participants will be assigned to receive navigation services(NS). Those who do not complete the COVID-19 testing will again be randomized and some will be assigned to Critical Dialogue (CD)
  Interventions: Behavioral: Navigation Services; Behavioral: Critical Dialogue
- Referral/tested/brochure (Experimental): After initial randomization, some participants will be assigned to receive standard referral services. Those who complete the COVID-19 testing will again be randomized and some will receive a digital brochure.
  Interventions: Behavioral: Referral and Digital Brochure
- Referral/tested/brief counseling (Experimental): After initial randomization, some participants will be assigned to receive standard referral services. Those who complete the COVID-19 testing will again be randomized and some will be assigned to receive Brief Counseling (BC).
  Interventions: Behavioral: Brief Counseling
- Referral/not tested/brochure (Experimental): After initial randomization, some participants will be assigned to receive standard referral services. Those who do not complete the COVID-19 testing will again be randomized and some will receive a digital brochure.
  Interventions: Behavioral: Referral and Digital Brochure
- Referral/not tested/critical dialogue (Experimental): After initial randomization, some participants will be assigned to receive standard referral services. Those who do not complete the COVID-19 testing will again be randomized and some will be assigned to Critical Dialogue (CD).
  Interventions: Behavioral: Critical Dialogue

INTERVENTIONS:
Behavioral: Navigation Services — Navigation services include assessment and support with service referrals. Each participant will meet with a peer navigator in person or on Zoom Conferencing for 30 minutes to go over results from their social and health needs assessment that is retrieved from the baseline assessment. The navigator shares information about COVID-19, answers questions about testing, and makes referrals to other needed services
  Arms: Navigation/not tested/critical dialogue; Navigation/not tested/navigation services; Navigation/tested/brief counseling; Navigation/tested/navigation services
Behavioral: Brief Counseling — Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
  Arms: Navigation/tested/brief counseling; Referral/tested/brief counseling
Behavioral: Critical Dialogue — Critical Dialogue includes three one-hour-long, open-group-sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.
  Arms: Navigation/not tested/critical dialogue; Referral/not tested/critical dialogue
Behavioral: Referral and Digital Brochure — Referral will consist of a five-minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing IL recommendations is e-mailed or texted to participants.
  Arms: Referral/not tested/brochure; Referral/tested/brochure

SUMMARY:
This study tests an adaptation of the HIV Continuum of Prevention, Care, and Treatment Framework (CoPCT) for use in tracking COVID-19 testing and follow-up in a medically and socially vulnerable population. This study uses an integrated research collaborative framework that facilitates dialogue among researchers, community members, and service providers as a tool for optimizing the adaptive intervention and will take place at the Comprehensive Behavioral Health Center (CCHC).

DETAILED DESCRIPTION:
This study will use the Multiphase Optimization Strategy (MOST) to optimize an adaptive intervention that successfully navigates COVID-19 medically or socially vulnerable people through a continuum of prevention, care and treatment (CoPCT) modeled on the HIV CoPCT. The COVID-19 CoPCT starts with testing and continues with successful adherence to prevention or treatment guidelines to help prevent and/or treat COVID-19. The study will assess the effectiveness of Navigation Services compared to referrals in increasing COVID-19 testing and Brief Counseling in increasing adherence to the State of IL recommendations for COVID-19 prevention and treatment. The study will also examine the effect of Critical Dialogue on testing behavior among people who decline to be tested for COVID-19. The investigators will develop decision rules about what evidence-based-interventions work best for what types of people (e.g., those who test right away, versus decliners) and in what period of the COVID-19 continuum. Finally, the study will shed light on factors associated with testing and adherence to IL recommendations. Investigators will follow Community Based Participatory Research principles in implementing a sequential, multiple assignment randomized trial (SMART) design. Adjusting for possible 15% loss to follow-up, a total sample of 548 people who are medically and socially vulnerable to infection and poor outcomes with COVID-19 will be enrolled as the intent-to treat-sample. The investigators are confident that they can recruit this sample in St. Clair County, IL based on their previous experience and because the research team has established relationships with other service agencies in the community from which, in addition to CBHC, research participants will be drawn. The primary outcome is completion of the COVID-19 test within one week of the first intervention session. The study will include 3 stages in which participants will be randomized to one of two possible interventions as follows:

1. Eligible and consenting participants will be randomized to receive the first-stage intervention: Navigation Services (NS) or standard services (referral to testing and IL digital information brochure after testing). The primary outcome is completion of the COVID-19 test within one week of the intervention session.
2. Those who get tested will be randomized to receive the second-stage intervention: continue with NS or standard treatment or switch to Brief Counseling (BC). The outcome will be adherence to IL recommendations. For those testing positive, adherence means engaging in a 14-day quarantine, receiving medical care as needed and contact tracing. For those testing negative, adherence means social distancing and wearing masks.
3. Those who do not get tested will be randomized into their second-stage intervention to continue with NS or digital brochure or switch to Critical Dialogue (CD). The outcome will be completing COVID-19 testing within 1 week of the second stage intervention session. Those who complete the testing will then be randomized to either continue with NS or digital brochure or switch to BC. Those who do not get tested will be randomized to continued NS or digital brochure or switch to CD. The outcome will be adherence to NJ recommendations, as defined above. All variables will be measured using standardized measures selected from the National Institutes of Health (NIH) PhenX Toolkit.

For the primary aim of comparing effects of Navigation Services versus referral on testing behavior and IL recommendations adherence, using standard sample size formula for difference of two proportions, a total sample size of 466 subjects is needed to have 80% power at α=0.05 to detect a 10% difference in proportions, assuming 70% in the referral group will complete testing and adhere to specific IL recommendations. The 466 sample size has 85% to detect a difference of 15% in adherence rates to IL recommendations between two interventions.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* having high risk to contract COVID or develop related complications
* able to speak English
* able and willing to provide informed consent.

Exclusion Criteria:

* under 18 years of age
* not at high risk to contract COVID or develop related complications
* unable to speak English
* unable and unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Behavioral Health Center, East Saint Louis, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data can be shared upon request for research purposes and under a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon request after the study is complete
Access Criteria: Must sign a data sharing agreement

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited into the study at the Comprehensive Behavioral Health Center (CBHC), one of southern Illinois' largest and most comprehensive behavioral health providers.
Groups:
- Stage 1: Navigation: Participants in this arm were randomized to receive Navigation Services for Stage 1
- Stage 2 Navigation Followed by Navigation: Participants in this arm were first randomized to receive Navigation Services in Stage 1 and then were randomized again to receive Navigation Services in Stage 2 Navigation Services: Navigation services include assessment and support with service referrals. Each participant will meet with a peer navigator in person or on Zoom Conferencing for 30 minutes to go over results from their social and health needs assessment that is retrieved from the baseline assessment. The navigator shares information about COVID-19, answers questions about testing, and makes referrals to other needed services
- Stage 2: Navigation Followed by Brief Counseling: Participants in this arm were randomized into Navigation Services in Stage 1 then randomized into Brief Counseling in Stage 2.
  Brief Counseling: Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
- Stage 2: Navigation Followed by Critical Dialogue: Participants in this arm were first randomized to receive Navigation Services in Stage 1 then randomized to receive Critical Dialogue in Stage 2.
  Critical Dialogue: Critical Dialogue includes three one-hour-long, open-group- sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.
- Stage 1: Brochure: Participants in this group were randomized to receive a digital brochure in Stage 1.
  Referral and Digital Brochure: Referral will consist of a five- minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is e-mailed or texted to participants.
- Stage 2: Brochure Followed by Brochure: Participants in this group were randomized to receive a brochure in Stage 1 and randomized to receive a brochure in Stage 2.
  Referral and Digital Brochure: Referral will consist of a five- minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is e-mailed or texted to participants.
- Stage 2: Brochure Followed by Brief Counseling: Participants in this group were randomized to receive a brochure in Stage 1 and randomized to receive Brief Counseling in Stage 2.
  Brief Counseling: Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention
- Stage 2: Brochure Followed by Critical Dialogue: Participants in this group were randomized to receive a Brochure in Stage 1 and randomized to receive Critical Dialogue in Stage 2.
  Critical Dialogue: Critical Dialogue includes three one-hour-long, open-group- sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.
Period: Stage 1: First Intervention
Arm/Group | Stage 1: Navigation | Stage 2 Navigation Followed by Navigation | Stage 2: Navigation Followed by Brief Counseling | Stage 2: Navigation Followed by Critical Dialogue | Stage 1: Brochure | Stage 2: Brochure Followed by Brochure | Stage 2: Brochure Followed by Brief Counseling | Stage 2: Brochure Followed by Critical Dialogue
Started | 278 | 0 | 0 | 0 | 276 | 0 | 0 | 0
Completed | 132 | 0 | 0 | 0 | 276 | 0 | 0 | 0
Not Completed | 146 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2: Second Intervention
Arm/Group | Stage 1: Navigation | Stage 2 Navigation Followed by Navigation | Stage 2: Navigation Followed by Brief Counseling | Stage 2: Navigation Followed by Critical Dialogue | Stage 1: Brochure | Stage 2: Brochure Followed by Brochure | Stage 2: Brochure Followed by Brief Counseling | Stage 2: Brochure Followed by Critical Dialogue
Started (5 participants were not randomized following Stage 1) | 0 | 141 | 10 | 126 | 0 | 140 | 6 | 126
Completed | 0 | 24 | 10 | 15 | 0 | 5 | 6 | 23
Not Completed | 0 | 117 | 0 | 111 | 0 | 135 | 0 | 103

BASELINE CHARACTERISTICS:
Groups:
- Navigation (Stage 1) + Navigation (Stage 2): Participants in this group were randomized in Stage 1 to receive Navigation Services and randomized to receive Navigation Services in Stage 2.
  Navigation Services: Navigation services include assessment and support with service referrals. Each participant will meet with a peer navigator in person or on Zoom Conferencing for 30 minutes to go over results from their social and health needs assessment that is retrieved from the baseline assessment. The navigator shares information about COVID-19, answers questions about testing, and makes referrals to other needed services
- Navigation (Stage 1) + Brief Counseling (Stage 2): Participants in this Group were randomized to receive Navigation services in Stage 1 and randomized to receive Brief Counseling in Stage 2.
  Brief Counseling: Brief Counseling is a 15-minute post- COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
- Navigation (Stage 1) + Critical Dialogue (Stage 2): Participants in this group were randomized to receive Navigation Services in Stage 1 and randomized to receive Critical Dialogue in Stage 2.
  Critical Dialogue: Critical Dialogue includes three one- hour-long, open- group-sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities
- Brochure (Stage 1) + Brochure (Stage 2): Participants in this group were randomized in stage 1 to receive a digital brochure and randomized to receive a digital brochure in Stage 2.
  Referral and Digital Brochure: Referral will consist of a five- minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is e-mailed or texted to participants.
- Brochure (Stage 1)+ Brief Counseling (Stage 2): Participants in this group were randomized in Stage 1 to receive a Brochure and were randomized to receive Brief Counseling in Stage 2.
  Brief Counseling: Brief Counseling is a 15-minute post- COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention.
- Brochure (Stage 1) + Critical Dialogue (Stage 2): Participants in this group were randomized to receive Navigation Services in Stage 1 and were randomized to receive Critical Dialogue in Stage 2.
  Critical Dialogue: Critical Dialogue includes three one- hour-long, open- group-sessions facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the NCCB to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.
- Not Randomized After Stage 1: Participants in this group were not randomized following Stage 1
- Total: Total of all reporting groups
Arm/Group | Navigation (Stage 1) + Navigation (Stage 2) | Navigation (Stage 1) + Brief Counseling (Stage 2) | Navigation (Stage 1) + Critical Dialogue (Stage 2) | Brochure (Stage 1) + Brochure (Stage 2) | Brochure (Stage 1)+ Brief Counseling (Stage 2) | Brochure (Stage 1) + Critical Dialogue (Stage 2) | Not Randomized After Stage 1 | Total
Number analyzed (Participants) | 141 | 10 | 126 | 140 | 6 | 126 | 5 | 554
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3
  Between 18 and 65 years | 134 | 10 | 119 | 133 | 5 | 118 | 5 | 524
  >=65 years | 7 | 0 | 6 | 6 | 1 | 7 | 0 | 27
Sex/Gender, Customized [Number; unit: participants]
  Female | 74 | 6 | 66 | 63 | 4 | 73 | 2 | 288
  Male | 60 | 4 | 54 | 73 | 1 | 48 | 3 | 243
  Unknown/Unreported | 7 | 0 | 6 | 4 | 1 | 5 | 0 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 0 | 6 | 2 | 1 | 3 | 1 | 20
  Not Hispanic or Latino | 121 | 8 | 106 | 123 | 5 | 108 | 4 | 475
  Unknown or Not Reported | 13 | 2 | 14 | 15 | 0 | 15 | 0 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 0 | 4 | 1 | 0 | 5 | 0 | 15
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 112 | 9 | 93 | 106 | 3 | 92 | 4 | 419
  White | 14 | 1 | 18 | 20 | 2 | 21 | 0 | 76
  More than one race | 1 | 0 | 6 | 6 | 0 | 3 | 0 | 16
  Unknown or Not Reported | 9 | 0 | 5 | 6 | 1 | 4 | 1 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 141 | 10 | 126 | 140 | 6 | 126 | 5 | 554
COVID tested within previous 30 days [Count of Participants; unit: Participants] | 39 | 4 | 22 | 27 | 3 | 26 | 1 | 122

OUTCOME MEASURES:

1. Primary Outcome: Completion of COVID-19 Test
Description: Eligible and consenting participants will be randomized to receive the first-stage intervention: Navigation Services (NS) or standard services (referral to testing and IL digital information brochure after testing). The primary outcome is completion of the COVID-19 test within one week of the intervention session.
Time Frame: Within one week of the intervention session
Measure: Count of Participants; unit: Participants
Groups:
- Navigation (Stage 1): Participants in this group are randomized to receive Navigation Services in Stage 1.
  Navigation Services: Navigation services include assessment and support with service referrals. Each participant will meet with a peer navigator in person or on Zoom Conferencing for 30 minutes to go over results from their social and health needs assessment that is retrieved from the baseline assessment. The navigator shares information about COVID-19, answers questions about testing, and makes referrals to other needed services
- Brochure Only: After initial randomization, some participants will be assigned to receive standard referral services. Those who complete the COVID-19 testing will again be randomized and some will receive a digital brochure. Referral and Digital Brochure: Referral will consist of a five-minute phone call where an outreach worker offers participants information about COVID-19 testing and encourages them to get tested within one week. A digital brochure containing NJ recommendations is emailed or texted to participants.
Arm/Group | Navigation (Stage 1) | Brochure Only
Number analyzed (Participants) | 278 | 276
Participants | 72 | 60

2. Primary Outcome: Stage 2: Reported COVID Test in Last 30 Days at 6 Months Post Baseline
Description: For the second stage intervention, the primary outcome is self-reported completion of COVID-19 test in the past 30 days at the follow up completed 6 months after baseline. Study participants were asked whether they had completed a COVID-19 test in the past 30 days.
Time Frame: Stage 2: 6 months post baseline (4th follow up visit)
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation (Stage 1) + Navigation (Stage 2) | Navigation (Stage 1) + Brief Counseling (Stage 2) | Navigation (Stage 1) + Critical Dialogue (Stage 2) | Brochure (Stage 1) + Brochure (Stage 2) | Brochure (Stage 1)+ Brief Counseling (Stage 2) | Brochure (Stage 1) + Critical Dialogue (Stage 2)
Number analyzed (Participants) | 141 | 10 | 126 | 140 | 6 | 126
Participants | 39 | 4 | 23 | 27 | 3 | 26

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline through follow up sessions (6 months)
Groups:
- Not Randomized After Stage 1: Participants in this group were not randomized after Stage 1.
Arm/Group | Stage 1: Navigation | Stage 2 Navigation Followed by Navigation | Stage 2: Navigation Followed by Brief Counseling | Stage 2: Navigation Followed by Critical Dialogue | Stage 1: Brochure | Stage 2: Brochure Followed by Brochure | Stage 2: Brochure Followed by Brief Counseling | Stage 2: Brochure Followed by Critical Dialogue | Not Randomized After Stage 1
All-Cause Mortality (participants affected / at risk) | 0/278 | 0/138 | 0/10 | 0/126 | 0/273 | 0/128 | 0/6 | 0/122 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/278 | 0/138 | 0/10 | 0/126 | 0/273 | 0/128 | 0/6 | 0/122 | 0/5
Other Adverse Events (participants affected / at risk) | 0/278 | 0/138 | 0/10 | 0/126 | 0/273 | 0/128 | 0/6 | 0/122 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/43/NCT05305443/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT05305443/SAP_001.pdf